CLINICAL TRIAL: NCT00992199
Title: Randomized Controlled Trials on Adjuvant Intraperitoneal Chemotherapy for Resectable Local Advanced Gastric Cancer
Acronym: IPchemo-AGC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Haiyi Guo, Fudan University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IP chemo-AGC
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Gastric Cancer
Keywords: intraperitoneal chemotherapy; cisplatin; fluorouracil; advanced gastric cancer
MeSH Terms: interventions — CF regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control arm (No Intervention): adjuvant intravenous system chemotherapy
- IP Chemo arm (Experimental): adjuvant system intravenous chemotherapy combined with adjuvant intraperitoneal chemotherapy
  Interventions: Drug: cisplatin, Fluorouracil

INTERVENTIONS:
Drug: cisplatin, Fluorouracil — cisplatin,60mg,plus 5-Fu,1.0g,intraperitoneal administration,once a week for 3 times
  Other Names: DDP,5-Fu
  Arms: IP Chemo arm

SUMMARY:
Gastric cancer is the leading cause of death from a intestinal tract cancer in China.In most cases, the high death rate is due to tumor that has spread beyond the gastric cancer at the time of diagnosis. In China, the standard chemotherapy for the initial treatment of gastric cancer is a combination of a platinum analogue with 5-Fu.With modern surgical interventions and contemporary chemotherapy, most patients attain better clinical remission.The majority of them, however, will eventually have a relapse and die of the disease.

The peritoneal cavity is the principal site of disease in gastric cancer.Although the intensity of intravenous chemotherapy is limited mainly by myelotoxicity, several active drugs can be administered directly into the peritoneal cavity. The rationale for intraperitoneal therapy in gastric cancer is that the peritoneum, the predominant site of tumor, receives sustained exposure to high concentrations of antitumor agents while normal tissues, such as the bone marrow, are relatively spared.

The investigators conducted this trial to investigate the efficacy and safety of intraperitoneal chemotherapy in advanced gastric cancer.

DETAILED DESCRIPTION:
To investigate efficacy and safety of intraperitoneal chemotherapy as part of adjuvant treatment for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

* Histologically confirmed primary adenocarcinoma of the stomach
* 3-4weeks after radical operation for gastric cancer
* Stage of the gastric cancer was T3-4NxM0

PATIENT CHARACTERISTICS:

* Age: 18 - 70years old

Life expectancy:

* Longer than 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 80*10^12/mm3

Hepatic:

- AST no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy and radiotherapy were not allowed
* No other concurrent chemotherapy

Radiotherapy:

* Locally radiotherapy for local disease of advanced gastric cancer during adjuvant treatment was allowed

Surgery:

* See Disease Characteristics
* Prior surgery for gastric cancer was necessary

Exclusion Criteria:

* Haven't recovery from operation or complication of operation
* With the following risk factors: Uncontrolled or severe cardiovascular disease (e.g., myocardial infarction within the past 6 months, congestive heart failure treated with medications, or uncontrolled hypertension)
* Pregnant or nursing
* Other currently active malignancy except nonmelanoma skin cancer
* Uncontrolled or severe bleeding,diarrhea,intestinal obstruction,adhesion of intestine
* metastasis before enrollment
* Received other chemotherapy or radiotherapy after operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Metastasis in Peritoneum and peritoneal cavity | 1 year

SECONDARY OUTCOMES:
Liver metastasis | 1 year
Refraction-free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — member of Fudan University Cancer Hospital
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China